CLINICAL TRIAL: NCT01557842
Title: Early Ablation Therapy for the Treatment of Ischemic Ventricular Tachycardia in Patients With Implantable Cardioverter Defibrillators
Acronym: ASPIRE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASPIRE
Record Dates: First submitted 2012-03-16; First posted 2012-03-20 (Estimated); Results first posted 2015-01-01 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2017-05

CONDITIONS: Ventricular Tachycardia; Ischemic
Keywords: Ischemic; Ventricular Tachycardia; Implantable Cardioverter Defibrillators; Antiarrhythmic Drug Therapy; Ablation; Electrophysiology
MeSH Terms: conditions — Tachycardia, Ventricular; Ischemia | interventions — Catheter Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Group (Active Comparator): This group receives radiofrequency catheter ablation and drug treatment.
  Interventions: Device: Catheter Ablation
- Control Group (Experimental): This group receives only drug treatment.
  Interventions: Drug: Drug Treatment

INTERVENTIONS:
Drug: Drug Treatment — Class I and III antiarrhythmic drug treatment.
  Arms: Control Group
Device: Catheter Ablation — Radiofrequency catheter ablation and Class I and III antiarrhythmic drug treatment.
  Arms: Treatment Group

SUMMARY:
The purpose of this study is to determine if early ablation (i.e., ablation of ventricular tachycardia in patients with infrequent VT episodes) is more effective than medical therapy alone for the treatment of ischemic ventricular tachycardia in patients with Implantable Cardioverter Defibrillators (ICDs) who continue to have episodes of ventricular tachycardia despite drug therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be drug refractory on Class I-IV AADs (i.e., having VT episodes despite drug therapy)

   a. Subject must be on at least one AAD at time of enrollment
2. Qualifying episode must be sustained, monomorphic Ventricular Tachycardia post myocardial infarction
3. ICD implanted
4. 1 to 3 sustained monomorphic VT episodes requiring appropriate therapy within the previous six (6) months as determined by the investigator
5. History of myocardial infarction documented by the development of pathological Q waves with or without symptoms, imaging evidence of a region of loss of viable myocardium that is thinned and fails to contract in the absence of a nonischemic cause, or pathological findings of a healed or healing myocardial infarction
6. 18 years or older
7. Able and willing to comply with all pre- and follow-up testing and requirements
8. Signed Informed Consent Form

Exclusion Criteria:

1. Age < 18 years
2. Documented intra-atrial or ventricular thrombus or other abnormality on preablation echocardiogram
3. Patients with Incessant Ventricular Tachycardia (continuous sustained VTs that recur promptly despite repeated intervention for termination over several (≥ 3) hours)
4. Contraindication to anticoagulation
5. NYHA class IV
6. Left ventricular assist devices (LVADs) or other circulatory assist devices
7. Stroke as confirmed by plasma d-dimer levels or acute myocardial infarction as documented by electrocardiogram or cardiac imaging within the past three (3) months. (Note that a small cardiac enzyme release resulting from being in VT/shocks/etc. is not considered a myocardial infarction.)
8. Patients with active ischemia who are eligible for revascularization
9. Patients with idiopathic Ventricular Tachycardia or Ventricular Tachycardia of non-ischemic cause (such as nonischemic cardiomyopathy)
10. Other disease process likely to limit survival to less than 12 months
11. Serum creatinine of ≥ 2.5mg/dl
12. Thrombocytopenia or coagulopathy
13. Prior ablation for Ventricular Tachycardia
14. Women who are pregnant (as evidenced by pregnancy test if pre-menopausal)
15. Enrollment in an study evaluating an investigational device or drug
16. Unable or unwilling to comply with protocol requirements
17. Exclusively Polymorphic Ventricular Tachycardia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-06-01 (Actual); Primary Completion 2014-03-19 (Actual); Study Completion 2014-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Callans, MD, Study Chair — University of Pennsylvania; Francis Marchlinski, MD, Study Chair — University of Pennsylvania; Andrea Natale, MD, Study Chair — Texas Cardiac Arrhythmia Research Foundation; Vivek Reddy, MD, Study Chair — Icahn School of Medicine at Mount Sinai; David Wilber, MD, Study Chair — Loyola University
Locations (23):
- United States (23):
  - University of California, Los Angeles, Los Angeles, California
  - California Pacific Medical Center, San Francisco, California
  - San Francisco VA Medical Center, San Francisco, California
  - University of California, San Francisco, San Francisco, California
  - University of Colorado, Denver, Aurora, Colorado
  - Florida Hospital, Orlando, Florida
  - Loyola University Chicago, Maywood, Illinois
  - Central Baptist Hospital, Lexington, Kentucky
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Mount Sinai School of Medicine, New York, New York
  - Columbia University- New York Presbyterian Hospital, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
  - St. Luke's Medical Center, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first and the last subject were enrolled on July 9, 2012 and on January 30, 2014 respectively. All ASPIRE sites were notified that the study was terminated due to ongoing enrollment issues on March 10, 2014. A total of 21 US study sites were activated with 7 sites enrolling subjects. The last follow-up visit was completed on April 21, 2014.
Groups:
- Catheter Ablation Group: Subjects were randomly allocated to treatment in a 1:1 fashion. Subjects randomized to this arm were treated with ventricular tachycardia ablation using the NAVISTAR THERMOCOOL Catheter in conjunction with Class I and III anti-arrhythmic medical therapy. Determination of optimal medical therapy was at the discretion of the investigator.
- Drug Treatment Group: Subjects randomized to this arm were treated with Class I and III anti-arrhythmic medication alone. Determination of optimal medical therapy was at the discretion of the investigator.
Period: Overall Study
Arm/Group | Catheter Ablation Group | Drug Treatment Group
Started | 9 | 6
Completed | 0 | 0
Not Completed | 9 | 6
Not completed — Lost to Follow-up | 0 | 1
Not completed — Death | 1 | 0
Not completed — Lack of Efficacy | 0 | 1
Not completed — Not Meet Inclusion/Exclusion Criteria | 3 | 0
Not completed — Study Terminated by Sponsor | 3 | 4
Not completed — Not Ablated | 2 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | Catheter Ablation Group | Drug Treatment Group | Total
Number analyzed (Participants) | 9 | 6 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.0 (14.4) | 63.3 (6.1) | 66.1 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 8 | 6 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 2 | 0 | 2
  White | 7 | 5 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 6 | 15

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Who Had Hospitalization for Ventricular Tachycardia (VT) Related Causes/Events
Description: The hospital admission date must occur after completing the 1-month follow-up visit for the event to be considered an effectiveness failure.
Time Frame: From one month to 2 years follow up
Population: All enrolled subjects
Measure: Number; unit: percentage of participants
Arm/Group | Catheter Ablation Group | Drug Treatment Group
Number analyzed (Participants) | 9 | 6
percentage of participants | 0 | 16.67

2. Primary Outcome: Cardiac-related Death
Description: Subjects with cardiac-related death
Time Frame: 2 years follow up
Population: All enrolled subjects
Measure: Number; unit: percentage of participants
Arm/Group | Catheter Ablation Group | Drug Treatment Group
Number analyzed (Participants) | 9 | 6
percentage of participants | 0 | 0

ADVERSE EVENTS:
Time Frame: During the 3-year follow-up after the ablation procedure.
Arm/Group | Catheter Ablation Group | Drug Treatment Group
Serious Adverse Events (participants affected / at risk) | 3/9 | 4/6
Other Adverse Events (participants affected / at risk) | 3/9 | 3/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Catheter Ablation Group (N=9) | Drug Treatment Group (N=6)
Heart Failure (Cardiac disorders) | 0 (0) | 1 (2)
Congestive Heart Failure (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular Tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Deep Venous Thrombosis Distal (Vascular disorders) | 0 (0) | 1 (1)
Adenocarcinoma Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Catheter Ablation Group (N=9) | Drug Treatment Group (N=6)
Heart Failure (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular Fibrillation (Cardiac disorders) | 1 (3) | 0 (0)
Ventricular Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular Tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Intracardiac Thrombus (Cardiac disorders) | 0 (0) | 1 (1)
Chronotropic Incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Neurological Symptom (Nervous system disorders) | 0 (0) | 1 (1)
Medical Device Removal (Surgical and medical procedures) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Deep Venous Thrombosis NOS (Vascular disorders) | 0 (0) | 1 (1)
Pseudomonas Infection (Infections and infestations) | 0 (0) | 1 (1)
Obstructive Sleep Apnea Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Please note that this study was terminated early and only 15 subjects were enrolled. As a result the reported results might be unreliable (unmonitored) and limited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There IS an agreement between the Principal Investigator (PI)/Institution and the Sponsor (or its agents) that restricts the PI's rights to discuss, present or publish trial results after the trial is completed. Please contact Biosense Webster, Inc. for additional information.